CLINICAL TRIAL: NCT04676503
Title: Vaginal and Rectal Colonization of Lactobacillus Crispatus NTCVAG04 Following Oral Administration in Patients With History of Vaginitis/Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NTC srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTCVAG04_02-2018
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Vaginitis; Vaginosis
MeSH Terms: conditions — Vaginitis; Vaginal Diseases

STUDY DESIGN:
Intervention Model Description: Open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Arm - Biovaginil 480 mg capsules (Experimental): All patients will be treated with 1 capsule/day of BIOVAGINIL for two treatment cycles of 14 days each.
  Interventions: Dietary Supplement: BIOVAGINIL

INTERVENTIONS:
Dietary Supplement: BIOVAGINIL — Biovaginil is a notified food supplement formulated as 480 mg capsules. Each capsule contains Lactobacillus crispatus NTCVAG04 3 billion and Vitamin A 120 μg.

SUMMARY:
The purpose of this study is to identify the presence of L. Crispatus in the rectum and vagina after oral administration of BIOVAGINIL by searching for specific DNA of the bacterial strain, to evaluate the tolerability of BIOVAGINIL and evaluate the minimum duration of the oral administration necessary to determine the appearance of L. Crispatus.

DETAILED DESCRIPTION:
In fertile, premenopausal healthy women, the vaginal ecosystem is dominated by Lactobacillus spp., but a diverse array of other bacteria can be present in much lower numbers. Over 120 species of Lactobacillus have been identified and more than 20 species have been detected in the vagina. Molecular-based techniques have demonstrated that healthy vaginal microflora does not contain high numbers of many different species of Lactobacillus. Rather, one or two lactobacilli from a range of three or four species (mainly L. crispatus and L. iners but also L. jensenii and L. gasseri) are dominant, whereas other species are rare, lower in titer and tend to be novel phylotypes.

Vaginitis is defined as a spectrum of conditions that cause vaginal and sometimes vulvar symptoms such as itching, burning, irritation, odor and vaginal discharge. Infection is the most common cause of vaginitis, including bacterial vaginosis (BV), vulvovaginal candidiasis and trichomoniasis. Bacterial vaginosis is a very common microbiological disturbance of the vaginal environment in adult women and is characterized by a depletion of lactobacilli in favor of an overgrowth of anaerobic bacteria. Colonization by L. crispatus or L. jensenii is associated with a lower frequency of bacterial vaginosis, and L. crispatus is strongly correlated with the absence of BV, low pH, negative whiff test, absence of clue cells and normal vaginal discharge.

Although antibiotic treatment of BV is strongly recommended, attempts at improving the efficacy of therapy are still a matter of debate. In fact, antimicrobial treatment of urogenital infections is not always effective, and problems remain due to bacterial and yeast resistance, recurrent infections and side effects. Alternative remedies are thus of interest and many studies have provided evidence of the beneficial functions of the human microbiota and prompted the selection of bacterial strains with health-promoting capacities for the treatment of conditions in which the microbiota, or its optimal functioning, is altered. The rationale for the use of probiotics in women is based on the genitourinary regulatory role played by the healthy vaginal microbiota and the need for restoration of this microbial ecosystem after insult.

Until today, the most common way of delivering probiotic lactobacilli was the administration of vaginal suppositories.However, this route will no longer be acceptable as products containing probiotics (live microorganisms) are not admissible as medical devices as per European Medical Device Regulation (EU) 2017/245. Oral administration therefore represents an alternative and more patient-friendly concept for the restitution of the normal vaginal microbiota. Indeed, several studies demonstrated the ability of rectal bacteria to move from the intestinal tract to the vagina. Moreover, it was recently demonstrated that the administration of a yoghurt containing Lactobacillus spp. including L.. crispatus in addition to antibiotic treatment may improve recovery rate and symptoms of BV and is well tolerated.

It is therefore reasonable to suppose that the oral administration of a food supplement containing an adequate concentration of a strain of L. crispatus, one of the predominant species, in the vaginal microbiota in asymptomatic women, may promote the re-colonization of the vaginal environment. Since this species is so representative and crucial in maintaining a healthy vaginal environment, we believe that it is of utter importance to understand its activity to fully disclose its potential.

The aim of this pilot study is to investigate the presence of Lactobacillus crispatus NTCVAG04 in the vagina after oral administration of BIOVAGINIL, a food supplement, as a precondition for the subsequent evaluation of the ability of NTCVAG04 to rebalance the local microbiota and promote healing and/or prevention of recurrences of vaginitis/vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18 years
* History of vaginitis/vaginosis
* Informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Need for treatment of vaginitis/vaginosis with any antibiotic drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Positivity for NTCVAG04 in rectal swabs collected at the end of the first treatment cycle. | At the end of the first cycle ( the cycle is 14 days - Visit 2 - 21st day (± 2) of the menstrual cycle in progress or following enrolment)
  A descriptive statistical analysis will be performed for the rectal swabs for NTCVAG04
Positivity for NTCVAG04 in rectal swabs collected at the end of the second treatment cycle. | At the end of the second treatment cycles (the cycle is 14 days - Visit 3 - 14th day (± 2) of the next menstrual cycle)
  A descriptive statistical analysis will be performed for the rectal swabs for NTCVAG04
Positivity for NTCVAG04 in vaginal swabs collected at the end of the first treatment cycle. | At the end of the first cycle (the cycle is 14 days - Visit 2 - 21st day (± 2) of the menstrual cycle in progress) or following enrolment
  A descriptive statistical analysis will be performed for the vaginal swabs for NTCVAG04
Positivity for NTCVAG04 in vaginal swabs collected at the end of the second treatment cycle. | At the end of the second treatment cycles (the cycle is 14 days - Visit 3 - 14th day (± 2) of the next menstrual cycle)
  A descriptive statistical analysis will be performed for the vaginal swabs for NTCVAG04

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 30 days
  Analysis of patients that reported an adverse events and analysis of number and type of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo De Leo, Principal Investigator — Ospedale Santa Maria alle Scotte
Locations (1):
- Azienda Ospedaliera Universitaria di Siena - Unità Operativa Semplice Ginecologia Endocrinologica Centro Sterilità di Coppia, Siena, SI, Italy